CLINICAL TRIAL: NCT05270655
Title: Effects of a Cognitive-behavioural Intervention on Anxiety, Depression and Quality of Life Among Ethiopian Children With Haematological Cancer Receiving Chemotherapy.
Brief Title: Cognitive-behavioural Intervention for Anxiety, Depression and Quality of Life Among Children Receiving Chemotherapy.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Tenaw Gualu MELESSE, Principal investigator, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CREC Ref. No.: 2021.729-T
Record Dates: First submitted 2022-02-27; First posted 2022-03-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Hematologic Malignancy; Anxiety; Depression; Quality of Life
Keywords: Cognitive Behavioral Therapy; Anxiety; Depression; Quality of life; Children; Hematologic Malignancy; Chemotherapy; Ethiopia
MeSH Terms: conditions — Hematologic Neoplasms; Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: Single-blind, multi-center, randomised controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive-behavioural intervention (Experimental): Five sessions of cognitive-behavioural intervention will be delivered on a weekly basis.
  Interventions: Other: Cognitive-behavioural intervention
- Usual care (No Intervention): Participants in the control group will receive the usual psychosocial care provided by the staff nurses. To offer them attention, a research assistant in each hospital will meet them every week for 30 minutes to ask them about treatment adherence and any other concerns. The parents will be invited to attend it if they want to do so. Each participant will be given an appointment slip and reminded with a phone call two days before the next appointment. For participants whose medical appointment is more than a week, the research will contact them via phone.

INTERVENTIONS:
Other: Cognitive-behavioural intervention — Participants in the experimental group will receive five sessions of cognitive-behavioural intervention. Each session will be conducted face-to-face for 30-35 minutes a week and supplemented by home-based practices. The first session is an introductory to cognitive-behavioural intervention, the second session includes identifying, evaluating and challenging maladaptive thoughts, beliefs and behaviour, the third session includes behavioural activation, the fourth session is deep breathing, and the last session includes treatment evaluation and relapse prevention. The interventions will be delivered before chemotherapy sessions to avoid fatigue and to increase the patient's engagement with the interventions. To establish a strong therapeutic alliance and enhance intervention delivery and family support, parents will be invited to attend the introduction of the first session and the summary of each session (the last five minutes).
  Arms: Cognitive-behavioural intervention

SUMMARY:
The diagnosis and treatment of paediatric cancer is the most stressful experience for children and their families. Nearly all paediatric cancer patients are presented with at least one psychosocial problem, of which, anxiety and depression often coexist and are most frequently reported. Poorly managed anxiety and depression causes emotional and behavioural problems, impairs relationships and functioning, decreases adhere to treatment, increases the burden of symptoms and significantly impacts quality of life and prognosis. Despite the high rates and negative impacts of anxiety and depression in paediatric oncology, they are poorly managed. Thus, to mitigate the burden of anxiety, depression and impaired quality of life, an age-appropriate cognitive-behavioural intervention shows promise when incorporated with the existing pharmacologic interventions.

This study aims to test how effective cognitive-behavioural intervention is to improve anxiety, depression and quality of life of children during chemotherapy.

The study will be conducted in two hospitals in Ethiopia and include 8-18-year-old children with haematological cancer receiving chemotherapy, able to communicate with the local language, Amharic, able to provide parental consent and child assent, and without history of developmental, psychological, psychiatric, hearing or speech problems.

The study will enroll up to 80 participants and randomise them into two groups, one group will receive a cognitive-behavioural intervention and the the other group will receive the usual psychosocial care provided by staff nurses. Participants in the cognitive-behavioural intervention group will receive five sessions of individual face to face cognitive-behavioural intervention. Each session will last approximately 30-35 minutes a week and supplemented by home-based practices. This study will use different intervention delivery strategies including psychoeducation, guided discovery or Socratic questioning, discussion, drawing, painting or writing, and play depending on the content of each session and maturity of the child.

The levels of anxiety, depression and quality of life will be measured before the intervention, after the intervention and one month after completion of the intervention in both groups.

DETAILED DESCRIPTION:
The application of cognitive-behavioural therapy (CBT) has been used for the management of anxiety and depression. Nowadays, evidence suggests that CBT has promising effects on improving psychological and health-related outcomes in children with cancer. CBT is a structured, and tailored psychotherapeutic intervention based on cognitive and behavioural approaches that helps to understand the underlying thoughts, feelings, and behaviours that mitigate between the course of the illness and the outcomes. It helps to modify dysfunctional thoughts and beliefs, reduce maladaptive behaviour and increase adaptive skills. It enables the patients to control their emotions and behaviour, to become their own therapist, to make the interventions sustainable and prevent relapse.

A systematic review and meta-analysis conducted shows cognitive-behavioural therapy has been used to manage stressful experiences including anxiety and depression among children during the course of cancer treatment. However, the studies included heterogenous participants across the cancer trajectory and employed different intervention delivery strategies. Additionally, majority of the included studies didn't specify the theory guiding the intervention development. Thus, developing and evaluating theory driven and age appropriate cognitive-behavioural intervention strategies for children undergoing chemotherapy is worthy of research. In this study, the Beck's cognitive model will be adopted to develop theory driven and age appropriate effective cognitive-behavioural intervention strategies for children receiving chemotherapy. The model was selected based on the results of the systematic review and other literatures on CBT.

The model describes the interactions among cognition, affection, and behaviour. Accordingly, it is not only the stressor but the perceptions and beliefs of the individual, and interpretation of a particular stressor that affect the emotional, physiological, and behavioural responses. Children with cancer usually have negative perceptions and thoughts about the self and others, the illness, and treatments such as chemotherapy. These distorted thoughts and negative strategies are often associated with emotional disturbances such as anxiety and depression. Cognitive-behavioural intervention helps to identify and modify distorted thought and behaviour, and develop cognitive and behavioural adaptations to improve emotional and behavioural responses. Cognitive adaptation is mainly achieved through cognitive restructuring such as identifying and challenging distorted thoughts and misinterpretations and developing coping strategies. Behavioural adaptation is largely achieved through behavioural activation such as identifying and introducing joyful activities. Changes in cognitive processes and developing adaptive behavioural activities increases coping strategies and reduces anxiety and depression symptoms, increase psychosocial functioning and quality of life due to improvement in stressful symptoms.

This study aims to evaluate the effects of a theory-based cognitive behavioural-intervention on anxiety, depression and quality of life among Ethiopian children with haematological cancer receiving chemotherapy.

In this study, it is hypothesised that when compared to the control group, participants receiving a cognitive-behavioural intervention will have;

1. Significantly decreased anxiety at the end of the intervention
2. Significantly decreased depression at the end of the intervention
3. Significantly increased quality of life at the end of the intervention

ELIGIBILITY:
Inclusion Criteria:

1. 8 to 18-year-old children
2. Diagnosed with haematological cancer
3. Receiving chemotherapy
4. Able to communicate (speak, read and write) with the local language, Amharic
5. Able to provide written parental consent and oral child assent

Exclusion Criteria:

1. Have a history of developmental problems, psychological or psychiatric illness
2. Unable to collaborate in the study due to acute illness
3. Have hearing or speech problems

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 76 (Actual)
Dates: Start 2022-04-12 (Actual); Primary Completion 2022-10-20 (Actual); Study Completion 2022-10-20 (Actual)

PRIMARY OUTCOMES:
Change in anxiety level | At three time points; before the intervention (T0, baseline), immediately after the intervention (T1, at 6 weeks) and one month after completion of the intervention (T2, at 10 weeks)
  Anxiety and depression will be assessed using a self-report 25-items (15-items for anxiety and 10-items for depression) Revised Child Anxiety and Depression Scale (RCADS). Each item will be rated on a four-point Likert scale (0-3) and the total score will be calculated by converting the row scores into T-scores. T scores of ≥65 to 70 and ≥ 70 show borderline clinical threshold and above clinical threshold respectively. The higher anxiety sub-scale score refers higher anxiety.

SECONDARY OUTCOMES:
Change in depression level | At three time points; before the intervention (T0, baseline), immediately after the intervention (T1, at 6 weeks) and one month after completion of the intervention (T2, at 10 weeks)
  A self-report 25-items items Revised Child Anxiety and Depression Scale (RCADS) will be used to assess the level of depression. The higher depression sub-scale score refers to higher depression level.
Change in quality of life | At three time points; before the intervention (T0, baseline), immediately after the intervention (T1, at 6 weeks) and one month after completion of the intervention (T2, at 10 weeks)
  Quality of life will be assessed using a child-report Quality of Life Inventory Generic Core Score 4.0 (PedsQLTM 4.0 GCS) for ages (8-12 and 13-18). Each item will be scored on a five-point Likert scale (0-4). The total score will be calculated reversely scoring the 0-4 scale items and linearly transforming to 0-100. A higher score indicates higher quality of life.

OTHER OUTCOMES:
Satisfaction with cognitive-behavioural intervention | Immediately after the completion of the intervention (T1, at 6 weeks)
  As part of process evaluation, satisfaction with cognitive-behavioural intervention among participants in the experimental group will be assessed using four four-point Likert scale questions. The satisfaction scores range from 0 to16 and a higher score refers to higher satisfaction with cognitive-behavioural intervention.
Demographic characteristics | Immediately before the intervention (T0, at baseline)
  Demographic characteristics of the participants

CONTACTS AND LOCATIONS:
Overall Officials: Tenaw G Melesse, PhD (c), Principal Investigator — The Nethersole School of Nursing, Faculty of Medicine, The Chinese University of Hong Kong; Janita PC Chau, PhD, Study Chair — The Nethersole School of Nursing, Faculty of Medicine, The Chinese University of Hong Kong
Locations (2):
- Ethiopia (2):
  - Tikur Anbesa specialised hospital, Addis Ababa
  - University of Gondar specialised hospital, Gonder

IPD SHARING:
Plan to Share IPD: No
To ensure privacy and confidentiality of the participants, individual participant data will not be shared.

REFERENCES:
- [Background] Arslan FT, Basbakkal Z, Kantar M. Quality of life and chemotherapy-related symptoms of Turkish cancer children undergoing chemotherapy. Asian Pac J Cancer Prev. 2013;14(3):1761-8. doi: 10.7314/apjcp.2013.14.3.1761. PMID 23679270
- [Background] Flowers SR, Birnie KA. Procedural Preparation and Support as a Standard of Care in Pediatric Oncology. Pediatr Blood Cancer. 2015 Dec;62 Suppl 5:S694-723. doi: 10.1002/pbc.25813. PMID 26700922
- [Background] Hsiao HJ, Chen SH, Jaing TH, Yang CP, Chang TY, Li MY, Chiu CH, Huang JL. Psychosocial interventions for reduction of distress in children with leukemia during bone marrow aspiration and lumbar puncture. Pediatr Neonatol. 2019 Jun;60(3):278-284. doi: 10.1016/j.pedneo.2018.07.004. Epub 2018 Jul 21. PMID 30100518
- [Background] Hyslop S, Davis H, Duong N, Loves R, Schechter T, Tomlinson D, Tomlinson GA, Dupuis LL, Sung L. Symptom documentation and intervention provision for symptom control in children receiving cancer treatments. Eur J Cancer. 2019 Mar;109:120-128. doi: 10.1016/j.ejca.2019.01.002. Epub 2019 Feb 1. PMID 30716715
- [Background] Lawlor C, Sharma B, Khondoker M, Peters E, Kuipers E, Johns L. Service user satisfaction with cognitive behavioural therapy for psychosis: Associations with therapy outcomes and perceptions of the therapist. Br J Clin Psychol. 2017 Mar;56(1):84-102. doi: 10.1111/bjc.12122. Epub 2016 Dec 2. PMID 27910997
- [Background] Levine DR, Mandrell BN, Sykes A, Pritchard M, Gibson D, Symons HJ, Wendler D, Baker JN. Patients' and Parents' Needs, Attitudes, and Perceptions About Early Palliative Care Integration in Pediatric Oncology. JAMA Oncol. 2017 Sep 1;3(9):1214-1220. doi: 10.1001/jamaoncol.2017.0368. PMID 28278329
- [Background] Li HC, Williams PD, Lopez V, Chung JO, Chiu SY. Relationships among therapy-related symptoms, depressive symptoms, and quality of life in Chinese children hospitalized with cancer: an exploratory study. Cancer Nurs. 2013 Sep-Oct;36(5):346-54. doi: 10.1097/NCC.0b013e31824062ec. PMID 23059766
- [Background] Li R, Ma J, Chan Y, Yang Q, Zhang C. Symptom Clusters and Influencing Factors in Children With Acute Leukemia During Chemotherapy. Cancer Nurs. 2020 Sep/Oct;43(5):411-418. doi: 10.1097/NCC.0000000000000716. PMID 31107701
- [Background] Lopez-Rodriguez MM, Fernandez-Millan A, Ruiz-Fernandez MD, Dobarrio-Sanz I, Fernandez-Medina IM. New Technologies to Improve Pain, Anxiety and Depression in Children and Adolescents with Cancer: A Systematic Review. Int J Environ Res Public Health. 2020 May 19;17(10):3563. doi: 10.3390/ijerph17103563. PMID 32438762
- [Background] Pitman A, Suleman S, Hyde N, Hodgkiss A. Depression and anxiety in patients with cancer. BMJ. 2018 Apr 25;361:k1415. doi: 10.1136/bmj.k1415. No abstract available. PMID 29695476
- [Background] Rossberg JI, Evensen J, Dammen T, Wilberg T, Klungsoyr O, Jones M, Boen E, Egeland R, Breivik R, Lovgren A, Ulberg R. Mechanisms of change and heterogeneous treatment effects in psychodynamic and cognitive behavioural therapy for patients with depressive disorder: a randomized controlled trial. BMC Psychol. 2021 Jan 22;9(1):11. doi: 10.1186/s40359-021-00517-6. PMID 33482927
- [Background] Walubita M, Sikateyo B, Zulu JM. Challenges for health care providers, parents and patients who face a child hood cancer diagnosis in Zambia. BMC Health Serv Res. 2018 May 2;18(1):314. doi: 10.1186/s12913-018-3127-5. PMID 29720168
- [Background] Yardeni M, Abebe Campino G, Hasson-Ohayon I, Basel D, Hertz-Palmor N, Bursztyn S, Weisman H, Pessach IM, Toren A, Gothelf D. Trajectories and risk factors for anxiety and depression in children and adolescents with cancer: A 1-year follow-up. Cancer Med. 2021 Aug;10(16):5653-5660. doi: 10.1002/cam4.4100. Epub 2021 Jul 26. PMID 34309238
- [Background] Zahed G, Koohi F. Emotional and Behavioral Disorders in Pediatric Cancer Patients. Iran J Child Neurol. 2020 Winter;14(1):113-121. PMID 32021635
- [Background] Zhang P, Mo L, Torres J, Huang X. Effects of cognitive behavioral therapy on psychological adjustment in Chinese pediatric cancer patients receiving chemotherapy: A randomized trial. Medicine (Baltimore). 2019 Jul;98(27):e16319. doi: 10.1097/MD.0000000000016319. PMID 31277176
- [Derived] Melesse TG, Li WHC, Chau JPC, Yimer MA, Gidey AM, Yitayih S. Cognitive-Behavioral Intervention for Children With Hematological Cancer Receiving Chemotherapy: A Randomized Controlled Trial. Psychooncology. 2025 Jan;34(1):e70086. doi: 10.1002/pon.70086. PMID 39828642
- [Derived] Melesse TG, Chau JPC, Li WHC. Efficacy of a culturally tailored cognitive-behavioural intervention for Ethiopian children with haematological malignancies: study protocol for randomised controlled trial. Trials. 2022 Sep 27;23(1):811. doi: 10.1186/s13063-022-06768-x. PMID 36163030